CLINICAL TRIAL: NCT04579562
Title: Regional Epidemiology of COVID-19 and Acute Kidney Injury in England
Brief Title: Regional COVID Epidemiology in England (RECEDE)
Acronym: RECEDE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UHDB/2020/075
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 positive AKI
  Interventions: Other: No intervention
- COVID-19 positive no AKI
  Interventions: Other: No intervention
- COVID negative AKI
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is observational, non-interventional study

SUMMARY:
The COVID-19 pandemic has exposed the unwanted variation in outcomes as evidence by Public Health England's report on increased mortality in regions of the country. For example, UHDB, in East Midlands, has reported a high crude mortality as compared to other Trusts in the region.8 There may also have been variation in the incidence of complications of COVID-19 in the form of AKI, which may have influenced mortality. Variation in outcomes may be because of various factors - differing population demographics, underlying health conditions in the population, deprivation, physician preference and knowledge and ethnic diversity. Unwanted variation is care that is not consistent with a patient's preference or related to [their] underlying illness. It is important to understand the reason for unwanted variation in outcomes associated with COVID-19 to minimise patient harm and reduce morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

This study will have two work packages (WP). Work Package 1 (WP1): Regional epidemiology of COVID-19 in England All patients who are admitted to hospital with COVID-19 infection between 1st March 2020 and 30th June 2020 and who meet following criteria will be included

1. Diagnostic code for COVID-19 (U07.1) in any of the 20 diagnoses codes
2. Adult patients greater or equal to 18 years of age.

Work Package 2 (WP2): Epidemiology of COVID-19 associated AKI in England All patients who are admitted to hospital with acute kidney injury (AKI) between 1st March 2020 and 30th June 2020 and who meet following criteria will be included

1. Diagnostic code for AKI (N17) in any of the 20 diagnoses codes
2. Adult patients greater or equal to 18 years of age.

Exclusion Criteria:

WP1:

The following patients will be excluded from the study

1. Patients not admitted to the hospital
2. Paediatric patients < 18 years of age

WP2:

The following patients will be excluded from the study

1. Patients not admitted to the hospital
2. Paediatric patients < 18 years of age
3. Patients on chronic maintenance haemodialysis or peritoneal dialysis

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will use analysis of all admitted patients in the past in England between 1st March 2020 and 30th June 2020 from the Hospital Episode Statistics (HES), a data warehouse containing details of all admissions at NHS hospitals in England. This design will help to analyse large number of AKI patients in short time-span so as to cascade the learning in timely fashion. HES collects a detailed record for each admitted patient care delivered in England, either by NHS hospitals. In each patient record, there are specific codes for additional diagnosis, or operations. We will extract all patients with diagnosis of COVID-19 by ICD-10 code of U07.1 and AKI as identified by ICD-10 code of N17 in any of the 20 diagnostic codes during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  In-hospital all cause mortality in patients with acute kidney injury and COVID-19
acute kidney injury | 30 days
  Incidence of acute kidney injury in patients with COVID-19

SECONDARY OUTCOMES:
Mechanical ventilation | 30 days
  Need for mechanical ventilation in patients with COVID-19

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 6 months

REFERENCES:
- [Derived] Kolhe NV, Fluck R, Taal M. Effect of COVID-19 with or without acute kidney injury on inpatient mortality in England: a national observational study using administrative data. BMJ Open. 2025 Mar 15;15(3):e095020. doi: 10.1136/bmjopen-2024-095020. PMID 40090681
- [Derived] Kolhe NV, Fluck RJ, Taal MW. Regional variation of COVID-19 admissions, acute kidney injury and mortality in England - a national observational study using administrative data. BMC Infect Dis. 2024 Mar 22;24(1):346. doi: 10.1186/s12879-024-09210-6. PMID 38519921